CLINICAL TRIAL: NCT05568628
Title: Ultrasonography Screening for Breast Lesions During Pregnancy and Lactation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hebatallah Gamal Ahmed, resident doctor at sohag cancer institute, Sohag University
Other Study IDs: Soh-Med-22-09-01
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Preganat and Lactating Faemls
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lacating femals: screening of breast lesions in lactating female
  Interventions: Device: ultrasound
- pregnant: screening of breast lesions in pregnant female
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — screening of breast lesions by ultrasonography

SUMMARY:
All breast disorders found during pregnancy and lactation should be carefully evaluated. Most of them are benign e.g., lactating adenoma, galactocele, fibroadenoma or inflammatory disorders e.g., mastitis, abscess formation, granulomatous mastitis, but it is essential to exclude pregnancy-associated breast cancer (PABC), which is too often diagnosed late Ultrasound is the first line breast imaging technique during pregnancy and lactation as Development of alveoli during pregnancy might not occur symmetrically, and these can be felt as focal nodularities, or even feel similar to masses, any suspicion of a mass should be assessed with US . If US illustrates glandular tissue and this correlates with the examiner presumption, no further work-up needs to be done. However, if presence of a mass is highly assumed, further follow-up by mammography, MRI and biopsy, when necessary, must be performed

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and lactating women with or without complaining of breast pain or breast lump referred from Obstetric and Gynecological outpatient clinic or surgery outpatient clinic

Exclusion Criteria:

* Non pregnant, non-lactating females, females with previous breast surgery or breast mass lesions before pregnancy or lactation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: - Pregnant and lactating women with or without complaining of breast pain or breast lump referred from Obstetric and Gynecological outpatient clinic or surgery outpatient clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
percent of breast lesions in pregnant and lactating females' | 12 month
  percent of breast lesions in pregnant and lactating females'

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Langer A, Mohallem M, Berment H, Ferreira F, Gog A, Khalifa D, Nekka I, Cherel P. Breast lumps in pregnant women. Diagn Interv Imaging. 2015 Oct;96(10):1077-87. doi: 10.1016/j.diii.2015.07.005. Epub 2015 Sep 2. PMID 26341843
- [Background] Langer A, Mohallem M, Stevens D, Rouzier R, Lerebours F, Cherel P. A single-institution study of 117 pregnancy-associated breast cancers (PABC): Presentation, imaging, clinicopathological data and outcome. Diagn Interv Imaging. 2014 Apr;95(4):435-41. doi: 10.1016/j.diii.2013.12.021. Epub 2014 Jan 31. PMID 24485752
- [Background] Genin AS, De Rycke Y, Stevens D, Donnadieu A, Langer A, Rouzier R, Lerebours F. Association with pregnancy increases the risk of local recurrence but does not impact overall survival in breast cancer: A case-control study of 87 cases. Breast. 2016 Dec;30:222-227. doi: 10.1016/j.breast.2015.09.006. Epub 2015 Oct 9. PMID 26456897
- [Background] Parker S, Saettele M, Morgan M, Stein M, Winkler N. Spectrum of Pregnancy- and Lactation-related Benign Breast Findings. Curr Probl Diagn Radiol. 2017 Nov-Dec;46(6):432-440. doi: 10.1067/j.cpradiol.2016.12.013. Epub 2016 Dec 27. PMID 28189388